CLINICAL TRIAL: NCT03176693
Title: Randomized Controlled Trial of Preoperative Alpha Blockade for Pheochromocytoma
Brief Title: Preoperative Alpha Blockade for Pheochromocytoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Masha Livhits, Co-Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB#17-000048
Record Dates: First submitted 2017-05-31; First posted 2017-06-05 (Actual); Results first posted 2023-11-20 (Actual); Last update posted 2023-11-20 (Actual); Status verified 2023-11

CONDITIONS: Pheochromocytoma; Paraganglioma
MeSH Terms: conditions — Pheochromocytoma; Paraganglioma | interventions — Phenoxybenzamine; Doxazosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phenoxybenzamine (Active Comparator): 3-4 weeks prior to date of surgery, patient will start phenoxybenzamine 10mg PO twice daily. Phenoxybenzamine will then be titrated to a blood pressure <120/80 (sitting) with mild orthostatic hypotension (drop in systolic blood pressure by 20 points or diastolic blood pressure by 10 points from sitting to standing position); systolic blood pressure not less than 90 (standing).
  Interventions: Drug: Phenoxybenzamine
- Doxazosin (Experimental): 3-4 weeks prior to date of surgery, patient will start doxazosin 1 mg PO daily. Phenoxybenzamine will then be titrated to a blood pressure <120/80 (sitting) with mild orthostatic hypotension (drop in systolic blood pressure by 20 points or diastolic blood pressure by 10 points from sitting to standing position); systolic blood pressure not less than 90 (standing).
  Interventions: Drug: Doxazosin

INTERVENTIONS:
Drug: Phenoxybenzamine — Non-selective alpha blocker
  Other Names: Dibenzyline
  Arms: Phenoxybenzamine
Drug: Doxazosin — Selective alpha blocker
  Other Names: Cardura
  Arms: Doxazosin

SUMMARY:
Pheochromocytoma is a rare, catecholamine (ex. adrenaline) secreting tumor that requires preoperative alpha blockade to minimize intraoperative hemodynamic instability, thereby reducing intra- and postoperative morbidity and mortality. Phenoxybenzamine is a non-selective alpha blocker that is significantly more expensive and is associated with increased adverse effects in comparison with selective alpha blockers such as doxazosin. Retrospective studies show minimal differences in hemodynamic instability and no differences in postoperative morbidity and mortality between selective vs. non-selective alpha blockers. This study is a randomized controlled trial that will compare hemodynamic instability, morbidity, mortality, cost, and quality of life between patients blocked with phenoxybenzamine vs. doxazosin.

DETAILED DESCRIPTION:
Pheochromocytoma is a catecholamine (ex. adrenaline) secreting tumor for which the primary treatment is surgical resection. Due to the hormones secreted by the tumor, alpha receptors on peripheral blood vessels are activated, causing constriction of these blood vessels and dangerously high blood pressure. During resection of the tumor, the source of excess hormone secretion is abruptly removed, which can lead to life-threatening blood pressure fluctuations during surgery.

Alpha blockers are a class of medication that blocks the alpha receptor on blood vessels. Given preoperatively over a few weeks, these medications negate the effects of the excess hormones secreted by the pheochromocytoma, reducing the frequency and severity of dangerous blood pressure fluctuations intraoperatively and postoperatively. Preoperative alpha blockade is therefore critical to safely perform surgery to resect pheochromocytoma.

Phenoxybenzamine, a non-selective alpha blocker, is the most common medication used to alpha block patients prior to pheochromocytoma resection. However, due to increasing drug costs and increased side effects in comparison with selective alpha blockers, there is a renewed interest in studying alternatives to phenoxybenzamine.

Selective alpha blockers such as doxazosin are also commonly used to alpha block patients prior to pheochromocytoma resection. Selective alpha blockers are significantly less expensive and are associated with fewer side effects than phenoxybenzamine. Most retrospective studies comparing phenoxybenzamine with selective alpha blockers show no difference in intraoperative blood pressure fluctuations, morbidity, or mortality in pheochromocytoma resection. However, no prospective, randomized controlled trials comparing phenoxybenzamine to selective alpha blockers have been performed.

The purpose of our study is to analyze preoperative, intraoperative, and postoperative outcomes in patients randomized to receive phenoxybenzamine (non-selective) or doxazosin (selective) for alpha blockade prior to pheochromocytoma resection. Outcomes will include postoperative morbidity and mortality, intraoperative hemodynamic instability, quality of life, and cost.

ELIGIBILITY:
Inclusion Criteria:

* Adults with pheochromocytoma / paraganglioma undergoing surgical resection

Exclusion Criteria:

* Children < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2021-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Yeh, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Livingstone M, Duttchen K, Thompson J, Sunderani Z, Hawboldt G, Sarah Rose M, Pasieka J. Hemodynamic Stability During Pheochromocytoma Resection: Lessons Learned Over the Last Two Decades. Ann Surg Oncol. 2015 Dec;22(13):4175-80. doi: 10.1245/s10434-015-4519-y. Epub 2015 Mar 31. PMID 25822781
- [Background] Kesselheim AS, Avorn J, Sarpatwari A. The High Cost of Prescription Drugs in the United States: Origins and Prospects for Reform. JAMA. 2016 Aug 23-30;316(8):858-71. doi: 10.1001/jama.2016.11237. PMID 27552619
- [Result] Randle RW, Balentine CJ, Pitt SC, Schneider DF, Sippel RS. Selective Versus Non-selective alpha-Blockade Prior to Laparoscopic Adrenalectomy for Pheochromocytoma. Ann Surg Oncol. 2017 Jan;24(1):244-250. doi: 10.1245/s10434-016-5514-7. Epub 2016 Aug 25. PMID 27561909
- [Result] Kiernan CM, Du L, Chen X, Broome JT, Shi C, Peters MF, Solorzano CC. Predictors of hemodynamic instability during surgery for pheochromocytoma. Ann Surg Oncol. 2014 Nov;21(12):3865-71. doi: 10.1245/s10434-014-3847-7. Epub 2014 Jun 18. PMID 24939623
- [Result] Brunaud L, Boutami M, Nguyen-Thi PL, Finnerty B, Germain A, Weryha G, Fahey TJ 3rd, Mirallie E, Bresler L, Zarnegar R. Both preoperative alpha and calcium channel blockade impact intraoperative hemodynamic stability similarly in the management of pheochromocytoma. Surgery. 2014 Dec;156(6):1410-7; discussion1417-8. doi: 10.1016/j.surg.2014.08.022. Epub 2014 Nov 11. PMID 25456922
- [Result] Weingarten TN, Cata JP, O'Hara JF, Prybilla DJ, Pike TL, Thompson GB, Grant CS, Warner DO, Bravo E, Sprung J. Comparison of two preoperative medical management strategies for laparoscopic resection of pheochromocytoma. Urology. 2010 Aug;76(2):508.e6-11. doi: 10.1016/j.urology.2010.03.032. Epub 2010 May 23. PMID 20546874
- [Result] Prys-Roberts C, Farndon JR. Efficacy and safety of doxazosin for perioperative management of patients with pheochromocytoma. World J Surg. 2002 Aug;26(8):1037-42. doi: 10.1007/s00268-002-6667-z. Epub 2002 Jun 19. PMID 12192533

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 19 patients pretreated with phenoxybenzamine included for analysis: 15 historical patients who were pre-treated with phenoxybenzamine by their provider, 4 prospective randomized patients.
  20 patients pretreated with doxazosin included for analysis: 8 prospective randomized patients, 6 crossover patients (initially assigned phenoxybenzamine but elected to receive only doxazosin due to treatment cost), 6 prospective non-randomized patients
Period: Overall Study
Arm/Group | Phenoxybenzamine | Doxazosin
Started | 19 | 20
Completed | 19 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phenoxybenzamine | Doxazosin | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 52 [33 to 61] | 56 [35 to 68] | 54 [34 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 26
  Male | 7 | 6 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 16 | 15 | 31
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 10 | 16 | 26
  Black | 2 | 0 | 2
  Asian | 3 | 2 | 5
  Other/unknown | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 19 | 20 | 39

OUTCOME MEASURES:

1. Primary Outcome: Hemodynamic Instability
Description: Proportion of operative time outside target thresholds: SBP >180 or <80; DBP > 90; MAP>150 or <50; HR>90.
  Arterial line blood pressure measurements were extracted from the electronic medical record every 60 seconds.
Time Frame: Intraoperative, approximately 90 minutes
Measure: Median (Inter-Quartile Range); unit: percentage of total operative time
Arm/Group | Phenoxybenzamine | Doxazosin
Number analyzed (Participants) | 19 | 20
percentage of total operative time | 14 [5 to 34] | 13 [3 to 33]
Statistical Analysis 1: Comparison: Phenoxybenzamine vs Doxazosin; Null hypothesis: hemodynamic instability time will not differ between arms; Test type: Equivalence — A power analysis was calculated based on findings reported by Weingarten et al. of more frequent episodes of hypotension (defined as difference of mean systolic blood pressure <30% from baseline) in phenoxybenzamine compared with doxazosin (15.7% versus 5.1%). Using a standard deviation of 16 and 11 (derived from reported interquartile ranges, assuming normal distribution), respectively, to achieve 80% power using an alpha =.05, a total sample size of 56 patients was determined; p = .56, Wilcoxon (Mann-Whitney) — Threshold for statistical significance = 0.05

2. Secondary Outcome: Mortality
Description: Death within 30 days of surgery
Time Frame: 30 days postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Phenoxybenzamine | Doxazosin
Number analyzed (Participants) | 19 | 20
Participants | 0 | 0

3. Secondary Outcome: Daily Cost of Drug
Time Frame: Preoperative (2-3 weeks prior to surgery)
Measure: Median (Inter-Quartile Range); unit: Dollars
Arm/Group | Phenoxybenzamine | Doxazosin
Number analyzed (Participants) | 19 | 20
Dollars | 442.20 [323.44 to 634.58] | 5.06 [1.88 to 8.92]

4. Secondary Outcome: Quality of Life- Physical Functioning, Role Limitations Due to Physical Problems, Bodily Pain, General Health Perceptions, Vitality, Social Functioning, Role-limitations Due to Emotional Problems, and Mental Health
Description: Patients will take the SF-36 as well as a symptom survey describing the frequency and impact on their quality of life at several time points including prior to starting alpha blockade, immediately prior to surgery after being sufficiently blocked, and postoperatively at 30 days, 3 months, 6 months, and 1 year
Time Frame: From date of surgery (-2 to 3 weeks, -1 day, 30 days, 3 months, 6 months, 1 year)
Population: Due to staff turnover and COVID-19 restrictions, data was not collected or analyzed.
Arm/Group | Phenoxybenzamine | Doxazosin
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Morbidity as Assessed by Occurrence of Adverse Events
Description: Morbidity will be graded by Clavien Classification of adverse events
Time Frame: Postoperatively during inpatient stay and during readmissions up to 30 days postoperatively
Measure: Number; unit: events
Arm/Group | Phenoxybenzamine | Doxazosin
Number analyzed (Participants) | 19 | 20
events | 0 | 0

6. Secondary Outcome: Participants Admitted to Post-operative Intensive Care Unit (ICU)
Time Frame: up to 30 days post-surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Phenoxybenzamine | Doxazosin
Number analyzed (Participants) | 19 | 20
Participants | 2 | 1

ADVERSE EVENTS:
Time Frame: 30 days post-surgery
Arm/Group | Phenoxybenzamine | Doxazosin
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 0/19 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-15): https://cdn.clinicaltrials.gov/large-docs/93/NCT03176693/Prot_SAP_000.pdf